CLINICAL TRIAL: NCT05330845
Title: Interleukine 6 (IL6) Assay for Predicting Failure of Spontaneous Breathing in Patients With COVID-19 Acute Respiratory Distress Syndrome
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: end of recruitment period
Sponsor: Centre Hospitalier Henri Duffaut - Avignon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: COVIL6
Record Dates: First submitted 2022-04-07; First posted 2022-04-15 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: COVID-19 Acute Respiratory Distress Syndrome
Keywords: Interleukin-6; Acute Respiratory Distress Syndrome; COVID-19
MeSH Terms: conditions — Respiratory Distress Syndrome; COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with COVID-19 acute respiratory distress syndrome (Other): Patients with acute respiratory distress syndrome due to COVID-19 and requiring mechanical ventilation
  Interventions: Biological: IL6 assessment; Biological: CRP and PCT assessment

INTERVENTIONS:
Biological: IL6 assessment — Blood IL6 will be assessed during trial
Biological: CRP and PCT assessment — Blood CRP and PCT will be assessed during trial

SUMMARY:
In the current COVID-19 pandemic, many patients have an acute respiratory distress syndrome (ARDS). Among mechanisms related to COVID-19 acute respiratory distress syndrome, cytokine storm and secretion of IL-6 play a central role. ARDS management involves intubation for protective mechanical ventilation, deep sedation and curarisation.

During intensive care unit (ICU) hospitalization, improvement of hematosis induces a switch from a controlled ventilation mode to a withdrawal ventilation mode, such as Spontaneous Ventilation with Pressure Support (SP-PS) or Adaptative Support Ventilation (ASV). This step is essential prior to considering complete weaning from controlled ventilation and sometimes ends with a failure. In this case, deterioration of hematosis and/or ventilatory mechanics is observed.

At the same time as withdrawal failure, the investigators observed biological inflammatory rebound in some patients. Therefore, influence of inflammatory biological parameters, including IL-6, on withdrawal failure, needs to be investigated. To this end, the investigators decide to dose different inflammatory markers - such as IL6, C-Reactive Protein (CRP), Procalcitonin (PCT) - in patients with acute respiratory distress syndrome due to COVID-19, during standard of care. Indeed, in patients with acute respiratory distress syndrome not due to COVID-19, the increase in IL6 is a negative prognosis during medical first aid but also when the mechanical ventilation is withdrawn. In addition, IL6 rise is associated with poor prognosis for patients with COVID-19 and longer stays in intensive care.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years
* Patients with COVID-19 (positive COVID PCR)
* Use of intubation for mechanical ventilation

Exclusion Criteria:

* Use of Extracorporeal Membrane Oxygenation
* Treatment with Tocilizumab (anti-Il6)
* Pregnant woman
* Patients under protective administration or deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2021-08-05 (Actual); Primary Completion 2022-03-24 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Serum concentration of IL6 | Up to 72 hours after the start of respiratory weaning
  Change of blood IL6 concentration during switch from a controlled ventilation mode to a weaning ventilation mode in COVID-19 patients

SECONDARY OUTCOMES:
Serum concentration of CRP and PCT | Up to 48 hours after the start of respiratory weaning
  Change of blood CRP et PCT concentration during switch from a controlled ventilation mode to a weaning mode in COVID-19 patients
Pulmonary wedge pressure | Up to 48 hours after the start of respiratory weaning
  Change of pulmonary wedge pressure (in mmHg), respiratory rate (in breaths per minute), Fraction of inspired oxygen (FiO2, in percentage), Tidal Volume (in ml/kg) during switch from a controlled ventilation mode to a weaning mode in COVID-19 patients
Respiratory rate | Up to 48 hours after the start of respiratory weaning
  Change of respiratory rate (in breaths per minute) during switch from a controlled ventilation mode to a weaning mode in COVID-19 patients
Fraction of inspired oxygen | Up to 48 hours after the start of respiratory weaning
  Change of Fraction of inspired oxygen (FiO2, in percentage) during switch from a controlled ventilation mode to a weaning mode in COVID-19 patients
Tidal Volume | Up to 48 hours after the start of respiratory weaning
  Change of Tidal Volume (in ml/kg) during switch from a controlled ventilation mode to a weaning mode in COVID-19 patients
Days of mechanical ventilation | At the start of respiratory weaning
  Duration of mechanical ventilation (days)
Number of ventral decubitus | At the start of respiratory weaning
  Number of ventral decubitus during mechanical ventilation mode

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas POUSSARD, MD, Principal Investigator — Centre Hospitalier Henri Duffaut - Avignon; Estelle DELAUNAY, MD, Principal Investigator — Centre Hospitalier Henri Duffaut - Avignon
Locations (1):
- Centre Hospitalier Henri Duffaut, Avignon, Vaucluse, France

IPD SHARING:
Plan to Share IPD: No